CLINICAL TRIAL: NCT07203105
Title: GAINS Expert Guiding Technology to Coach Life Skill Teaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guiding Technologies Corporation (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R43MH130298-01 (NIH); 1R43MH130298-01 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: GAINS Expert Guiding Technology to Coach Life Skill Teaching
Keywords: Autism Spectrum Disorder; Technology; Behavior Intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAINS expert guiding technology to coach life skill teaching (Experimental)
  Interventions: Behavioral: GAINS expert guiding technology to coach life skill teaching

INTERVENTIONS:
Behavioral: GAINS expert guiding technology to coach life skill teaching — GAINS expert guiding technology to coach life skill teaching

SUMMARY:
Based on proven techniques in operant conditioning, the expert behavior guiding functionality in GAINS to teach life skills will be evaluated. Behavior practitioners will develop task analyses that break down complex life skills into simpler component steps and then enter these tasks into the GAINS system. In a similar way to navigation systems for drivers, GAINS will provide behavioral navigation for caregivers implementing ABA therapy programs. Using the GAINS app on a tablet or smartphone, caregivers will receive automatically updated visual and audio behavioral guidance, that includes what to do, when to do it, and detailed step-by-step guidance on how to execute ABA therapy programs.

ELIGIBILITY:
Inclusion Criteria:

* Only children ages 3 through 10 years who present with Autism Spectrum Disorder (ASD) will be recruited for this study.

Exclusion Criteria:

* No individuals will be excluded or included based on race, ethnicity, or gender

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Child independent life skill performance | 60 days
  The life skill steps (as determined by pre-treatment task analysis) the child performs without caregiver prompts divided by total life skill steps.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
SBIR Grant recipients are not required to share data.